CLINICAL TRIAL: NCT02513784
Title: Pilot Randomized Trial to Assess the Effects of an Antimicrobial Mouthwash on the Esophageal and Gastric Microbiome
Brief Title: Trial to Assess the Effects of an Antimicrobial Mouthwash on the Esophageal Microbiome
Acronym: Mouthwash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAP4553
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Adenocarcinoma; Barrett's Esophagus; Reflux Esophagitis
Keywords: Microbiome; Esophagus; Endoscopy; Mouthwash
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Barrett Esophagus; Esophagitis, Peptic | interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibacterial mouthwash (Experimental): Subjects will be randomized to twice daily chlorhexidine gluconate mouthwash for 21 days.
  Interventions: Drug: Chlorhexidine gluconate
- No intervention (No Intervention): Subjects will be randomized to no intervention for 21 days.

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Chlorhexidine gluconate is a germicidal mouthwash that reduces bacteria in the mouth.
  Other Names: Peridex
  Arms: Antibacterial mouthwash

SUMMARY:
This is a randomized, open-label pilot study to assess whether treatment with chlorhexidine mouthwash can alter the esophageal and gastric cardia microbiome

DETAILED DESCRIPTION:
Patients scheduled for upper endoscopy for clinical indications will be randomized to 3 weeks of either no treatment or use of twice daily chlorhexidine mouthwash leading up to the endoscopy. There will be 2-3 study visits, at Day 0 and Day 21, and for those subjects in the mouthwash arm, a final visit 1-2 weeks following the Day 21 visit. Subjects will be required to fast overnight prior to the visits on Days 0 and 21.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Scheduled for upper endoscopy for clinical indications
* No allergy or other contraindication to chlorhexidine

Exclusion Criteria:

* Use of proton pump inhibitors or H2 receptor antagonists within 1 month of enrollment. Acid suppressant medications raise the gastric pH and can dramatically alter the gastric and esophageal microbiome.
* History of upper gastrointestinal cancer
* History of histologically proven Barrett's esophagus
* History of antireflux or bariatric surgery, or other gastric or esophageal surgery
* Use of antimicrobial mouthwash within 1 month of enrollment
* Use of antibiotics or immunosuppressant medications within 3 months of enrollment
* Use of steroid inhalers or nasal sprays within 1 month of enrollment
* HIV or other immunosuppressed states or conditions (e.g. active malignancy)
* Pregnant or breast feeding
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian A. Abrams, MD, MS, Principal Investigator — Assistant Professor of Medicine and Epidemiology
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Annavajhala MK, May M, Compres G, Freedberg DE, Graham R, Stump S, Que J, Korem T, Uhlemann AC, Abrams JA. Relationship of the Esophageal Microbiome and Tissue Gene Expression and Links to the Oral Microbiome: A Randomized Clinical Trial. Clin Transl Gastroenterol. 2020 Dec;11(12):e00235. doi: 10.14309/ctg.0000000000000235. PMID 33512805
- See also: Clinical and Translational Gastroenterology: December 2020 - Volume 11 - Issue 12 — https://journals.lww.com/ctg/Fulltext/2020/12000/Relationship_of_the_Esophageal_Microbiome_and.13.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antibacterial Mouthwash | No Intervention
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antibacterial Mouthwash | No Intervention | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (12.9) | 51.2 (15.5) | 52.4 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20
Proton Pump Inhibitor (PPI) Use [Count of Participants; unit: Participants] | 5 | 5 | 10
Aspirin Use [Count of Participants; unit: Participants] | 4 | 4 | 8
Ever Smoker [Count of Participants; unit: Participants] | 3 | 3 | 6
Gastroesophageal Reflux Disease (GERD) History [Count of Participants; unit: Participants] | 7 | 9 | 16
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (6.0) | 31.2 (5.7) | 30.2 (5.8)
Waist to Hip Ratio (WHR) [Mean (Standard Deviation); unit: ratio] — Waist to Hip Ratio
  ratio | 0.94 (0.6) | 0.92 (0.8) | 0.93 (0.7)
Fat Intake [Mean (Standard Deviation); unit: % calories] | 35 (5.6) | 33.5 (2.6) | 34.3 (4.3)
Fiber intake [Mean (Standard Deviation); unit: gm/day] | 14.0 (3.8) | 13.6 (2.6) | 13.8 (3.2)
Indication for Upper Endoscopy (EGD) [Count of Participants; unit: Participants]
  Reflux symptoms | 5 | 4 | 9
  Abdominal pain | 2 | 2 | 4
  Dyspepsia | 1 | 2 | 3
  Other | 2 | 2 | 4
Endoscopic Findings [Count of Participants; unit: Participants]
  Reflux esophagitis | 2 | 3 | 5
  Varices | 1 | 0 | 1
  Normal esophagus | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Reduction of F. Nucleatum in Saliva
Description: Within individual change in relative abundance of F nucleatum in oral samples
Time Frame: 21 days
Population: Data was not collected and analyzed for F. Nucleatum in particular, instead an analysis was done for the microbiome composition across sample sites - oral swab, saliva and esophageal.
Arm/Group | Antibacterial Mouthwash | No Intervention
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Difference in Esophageal F. Nucleatum Between Experimental Group and no Intervention Group
Description: Comparison of relative abundance of esophageal F. nucleatum in the mouthwash group vs. the no intervention group.
Time Frame: 21 days
Population: as for outcome 1
Arm/Group | Antibacterial Mouthwash | No Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 days
Description: Participants were instructed to report any side effects of chlorhexidine. Tooth discoloration (a possible side effect of chlorhexidine use) was assessed by a dentist using photographs. The dentist was blinded to whether the images were from pre- or post-treatment.
Arm/Group | Antibacterial Mouthwash | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
There were no indications for repeated endoscopies, so the analysis of the esophagus was limited to a single point in time; relatively small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT02513784/Prot_SAP_000.pdf